CLINICAL TRIAL: NCT06913153
Title: Tianjin Diabetes and Health Cohort Study
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University (Other)
Responsible Party: Principal Investigator, Zhenqiang Song, Senior Researcher，Chu Hsien-I Memorial Hospital & Tianjin Institute of Endocrinology, Tianjin Medical University, Tianjin Medical University
Other Study IDs: TMUhMEC20250002
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus
Keywords: cohort study; diabets complication; etiology; clinical epidemiology; health economic evaluation
MeSH Terms: conditions — Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Diet

SUMMARY:
The goal of this observational study is to reveal the natural history of diabetes and the occurrence and development patterns of its complications, to evaluate the effectiveness of diabetes interventions, and to assess the health and medical burdens caused by diabetes in Tianjin, based on the medical records and health big data in Tianjin and correspondingly constructed diabetes-specific cohort.

DETAILED DESCRIPTION:
This study was conducted through the University-Enterprise Joint Laboratory for Diabetes Epidemiology Research at Tianjin Medical University. Retrospective and ongoing medical records and health big data from 396983 diabetes patients treated in secondary and tertiary hospitals in Tianjin between 2009 and 2024 were collected to establish a diabetes population cohort. Using advanced data mining techniques, multi-dimensional data including electronic health records (EHRs), medical imaging data, and wearable device metrics were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with diabetes
* Patients with three or more recorded visits
* The following information was complete at the first visit: age, sex, Blood Glucoseor ,glycated hemoglobin(HbA1c)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted through the University-Enterprise Joint Laboratory for Diabetes Epidemiology Research at Tianjin Medical University, China. Longitudinal multi-source health big data from 2009 to 2024 (encompassing 396,983 individuals with diabetes treated in secondary and tertiary healthcare facilities in Tianjin) were integrated to establish a representative diabetes population cohort.
Sampling Method: Probability Sample
Enrollment: 396983 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

IPD SHARING:
Plan to Share IPD: No
Access to raw datasets is restricted under legally binding agreements with the collaborating institutions, as these prohibit data sharing with third parties. However, de-identified aggregate findings, statistical summaries, or the study protocol can be made available upon reasonable request to the Principal Investigator (PI).

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is a real-world observational study and does not involve individual interventions or corresponding group assignment.
Groups:
- Cohort Comparising Patients With Diabetes: This dynamic cohort comparised 396983 diabetic patients who were enrolled in second- and tertiary-level hospitals in Tianjin during 2009-2024. All the participants had at least three medical visits.
Period: Overall Study
Arm/Group | Cohort Comparising Patients With Diabetes
Started | 396983
Completed | 396983
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Age, fasting blood glucose, and glycosylated hemoglobin were described using mean and standard deviation
Arm/Group | Cohort Comparising Patients With Diabetes
Number analyzed (Participants) | 396983
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181412
  Male | 215571
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 396983
  Race: Non-Asian | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 396983
medical history [Count of Participants; unit: Participants]
  The number of people with hypertension | 230484
  The number of people without hypertension | 166499
fasting glucose [Mean (Standard Deviation); unit: mmol/L] | 10.19 (4.01)
glycated hemoglobin [Mean (Standard Deviation); unit: %] | 7.43 (3.22)

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Complications
Description: Diabetic Complications: diabetic retinopathy,diabetic nephropathy,cerebral infarction,coronary artery disease The diagnosis of coronary artery disease is based on a comprehensive assessment of the degree of coronary artery stenosis and evidence of myocardial ischemia, taking into account risk factors and clinical symptoms, and exclusion of other similar diseases.
  The diagnostic criteria for diabetic nephropathy are history of diabetes: clear and long history of diabetes, Urine protein test:Urinary microalbumin excretion rate (UACR) is a key indicator for early diagnosis, with a normal value of less than 30mg/g, 30-300m Diagnosis of diabetic retinopathy by fundus examination. Diagnostic criteria for cerebral infarction are ICD codes or the doctor's diagnosis.
  Data collection through chart review, patient self-reporting, imaging
Time Frame: Baseline and week 520
Population: All the participants in the cohort are included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Coronary Artery Disease: The diagnosis of coronary artery disease is based on a comprehensive assessment of the degree of coronary artery stenosis and evidence of myocardial ischemia, taking into account risk factors and clinical symptoms, and exclusion of other similar diseases.The results for each outcome measure are presented in a table in which the columns represent the study's arms or comparison (analysis) groups and the rows present summary-level data. Each statistical analysis is similarly reported in a table that immediately follows the relevant outcome measure.
- Cerebral Infarction: Acute Onset and Symptomatic Features Sudden symptom onset, reaching peak within minutes to several hours, characterized by focal neurological deficits (e.g., unilateral limb weakness/numbness, speech disorders, facial asymmetry, visual disturbances, etc.).
  Symptom duration exceeds 24 hours, or imaging reveals a responsible ischemic lesion (e.g., CT hypodensity, MRI diffusion restriction).
  Imaging Evidence Head CT Scan: Excludes intracranial hemorrhage during the acute phase; low-density infarct lesions appear 24-48 hours post-onset.
  MRI (DWI Sequence): Highly sensitive, detecting ischemic lesions within minutes of symptom onset; preferred for early diagnosis.
  Vascular Imaging (CTA/MRA): Evaluates stenosis or occlusion of carotid/intracranial arteries, clarifying vascular lesion location and severity.
  Etiological Classification (at least one criterion must be met) Large Artery Atherosclerosis Type: Vascular stenosis >50% or occlusion with pathological atherosclerosis changes, excluding cardioembolic sources.
  Cardioembolic Type: Emboli of cardiac origin (e.g., atrial fibrillation, post-myocardial infarction mural thrombi) causing cerebral arterial occlusion, supported by ECG/echocardiographic evidence.
  Small Artery Occlusion Type (Lacunar Infarction): Infarct diameter <1.5-2.0 cm, predominantly in hypertensive patients, with mild symptoms and favorable prognosis.
- Diabetic Retinopathy: Diagnosis of diabetic retinopathy by fundus examination.
- Diabetic Nephropathy: The diagnostic criteria for diabetic nephropathy are history of diabetes: clear and long history of diabetes, Urine protein test:Urinary microalbumin excretion rate (UACR) is a key indicator for early diagnosis, with a normal value of less than 30mg/g, 30-300m
Arm/Group | Coronary Artery Disease | Cerebral Infarction | Diabetic Retinopathy | Diabetic Nephropathy
Number analyzed (Participants) | 396983 | 396983 | 396983 | 396983
Participants
  Patients presenting with any of the aforementioned clinical outcomes | 10263 | 97864 | 59029 | 69822
  Patients presenting without any of the aforementioned clinical outcomes | 386720 | 299119 | 337954 | 327161

2. Secondary Outcome: Glycemic Control
Description: Average level of glucose: including Glycated Hemoglobin (HbA1c), the mean of fasting glucose(FG) Glucose Variability: including standard deviation, coefficient of variation of HbA1c and FG.
Time Frame: baseline and week 520
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Mean Fasting Blood Glucose Level of the Population: Means and coefficients of variation of fasting blood glucose and glycosylated hemoglobin in the whole population
Arm/Group | Mean Fasting Blood Glucose Level of the Population
Number analyzed (Participants) | 396983
mmol/L | 8.7 (3.36)

3. Secondary Outcome: Death
Description: death from all cause, diabetes complications, and cancer.
Time Frame: baseline and week 520
Measure: Count of Participants; unit: Participants
Groups:
- All Cause: Refers to the sum of deaths from all causes during the study period, without distinguishing between specific causes of death
Arm/Group | All Cause
Number analyzed (Participants) | 396983
Participants
  Number of all-cause deaths | 21669
  Number of deaths not due to all causes | 375314

ADVERSE EVENTS:
Time Frame: This study is a real-world observational study and information on adverse events are not available .
Description: Deaths and adverse events were not assessed
Groups:
- Cohort Comparising Patients With Diabetes: This dynamic cohort comparised approximately 400,000 diabetic patients who were enrolled in second- and tertiary-level hospitals in Tianjin during 2009-2024. All the participants had at least three medical visits.
Arm/Group | Cohort Comparising Patients With Diabetes
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT06913153/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT06913153/SAP_001.pdf